CLINICAL TRIAL: NCT06651502
Title: Clinical and Radiographic Evaluations of Hiossen EK III NH Dental Implants
Brief Title: Efficacy of a Dental Implant System for Immediate Restoration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, David Kim, Associate Professor, Harvard Medical School (HMS and HSDM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-0702
Record Dates: First submitted 2024-09-30; First posted 2024-10-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Missing Teeth
Keywords: dental implant; immediate provisionalization
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- dental implant placement and immediate temporary restoration (Experimental): 1. pre-operative: comprehensive exam, standard-of-care x-rays, cone beam computed tomography (CBCT), dental optical scan
  2. intra-operative: dental implant placement and immediate provisionalization
  3. 4-week follow-up
  4. 12-week impression
  5. Delivery of final restoration
  6. follow-ups at 1 year and 2-year post-implant restoration
  Interventions: Device: dental implant placement and immediate provisionalization

INTERVENTIONS:
Device: dental implant placement and immediate provisionalization — dental implant placement and immediate temporization

SUMMARY:
The primary objective of this study is to observe the performance of an implant system with a new surface (EK III NH dental implants) over a period of two years. The implants will be placed in the upper and lower jaws of patients with missing teeth and immediately given a temporary restoration. The investigators will document the performance of the implants through regular dental check-ups and X-rays.

DETAILED DESCRIPTION:
Treating patients with missing teeth using dental implants is now a common and reliable approach in modern dentistry. Significant improvement has been made in implant shape design, implant surface optimization and surgical techniques to ensure predictable bonding between the titanium implants and bone (osseointegration). Modern implants are designed to be stable both immediately after placement (primary stability) and over time as they bond with the bone (secondary stability). Factors such as the quality and quantity of the patients' bone, the design of the implant, and the surgical technique used can all affect primary stability. The implant's secondary stability is affected by many of these same factors but has also been demonstrated to be influenced by other patient-related factors, including wound site blood supply, as well as the surface of the implants. Various surface treatments, like titanium plasma spraying, acid etching, hydroxyapatite coating, and sandblasting, have been developed to improve this bond (secondary stability). For instance, porous coatings can help by allowing the bone to grow into the implant, while hydroxyapatite coatings are biocompatible and encourage bone formation. Research has shown that different surface treatments can lead to different cellular responses, affecting how bone cells (osteoblasts) behave and develop around the implant.

In clinical practice, several methods are used to measure how stable an implant is immediately after placement, known as primary stability. These methods include measuring the insertion torque and using resonance frequency analysis (RFA). To assess secondary stability, or osseointegration, which refers to the long-term bonding of the implant to the bone, various techniques are used. These include RFA, mechanical disruption testing, and histomorphometric analysis. Additionally, changes in the bone level around the implant are commonly observed through X-rays as a non-invasive way to monitor the long-term success of dental implants. Human histological evidence of successfully osseointegrated implants is extremely rare in the literature because there are few opportunities to retrieve implants in humans.

Hiossen is a leading and rapidly growing implant manufacturer, with its systems used in over 70 countries. Recently, the company launched a new implant system called EK III NH. This system features a sand-blasted and acid-etched (SA) surface with a nano-hydroxyapatite (NH) coating. This special surface allows for faster bone healing and reduces the time before the implant can be loaded compared to other types of implant surfaces. The company's internal studies have shown that this surface treatment creates a very thin coating layer on the implant that is hydrophilic, meaning it attracts water, which improves the bonding process with 30% higher osseointegration than conventional SA surfaces. In addition, the new EK III NH system includes design improvements compared to the current ET SA implant system by the same company. New features include a buttress thread, 0.9 mm pitch, reverse helical cutting edge, and an improved internal hex connection, making the system easier to achieve good mechanical bonding immediately (primary stability) and easier to restore.

The investigators propose conducting a short-term clinical study to examine how well the bone around the EK III NH implants is maintained when they are immediately restored with a temporary crown. This study aims to assess the benefits of using the EK III NH implants in dental treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 20-80 years of age, who request dental implant treatment options to replace missing teeth as part of comprehensive dental care
* Subjects are willing to sign an informed consent, participate, and return for follow-up visits.
* Subjects without significant medical history and currently not on medications that might complicate the results

Exclusion Criteria:

* Subjects who do not meet all the inclusion criteria or will not cooperate with the protocol schedule.
* Subjects who received and failed a previously placed dental implant.
* Subjects who require a bone and soft tissue grafting procedure prior to or at the time of the implant placement.
* Subjects with significant untreated periodontal disease, caries, infection, or chronic inflammation in the oral cavity within two adjacent tooth positions of the clinical trial area.
* Subjects who have used nicotine-containing products within three weeks prior to surgery.
* Subjects who are insulin-dependent diabetic or if their Hgb1c levels > 6.5%.
* Subjects with a history of malignancy within the past five years (except for basal or squamous cell carcinoma of the skin or in situ cervical carcinoma).
* Subjects who are nursing or pregnant.
* Subjects who are presently taking medications (except estrogen/progesterone therapy) or those who are undergoing treatment that is known to affect bone turnover.
* Subjects with diseases affecting bone metabolism (excluding idiopathic osteoporosis).
* Subjects with a history of an autoimmune disease, documented allergy or multiple allergies to any component of the agents used in this study.
* Acutely infected defect site.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
radiographic crestal bone level | baseline, 12 weeks after implant, time of final restoration, 1-year post final restoration and 2-year post final restoration
  radiographs taken at baseline, 12 weeks following implant placement and at implant final restoration, 1 year after final restoration, and 2 years after final restoration will be analyzed for changes in the crestal bone level

SECONDARY OUTCOMES:
Implant Stability | at the time of implant placement
  Implant stability at the time of implant placement will be recorded using implant stability quotient. The usual range is between 50~80, the higher number indicates better stability.

CONTACTS AND LOCATIONS:
Overall Officials: David Kim, DDS, DMSc, Principal Investigator — Harvard School of Dental Medicine
Locations (1):
- Harvard Dental Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided